CLINICAL TRIAL: NCT00674895
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation for Control and Treatment of Parkinson's Disease.
Brief Title: Far Infrared Irradiation for Management and Treating of Parkinson's Disease (PD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-PD-CTP1
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Parkinson's Disease
Keywords: Idiopathic Parkinson's Disease; Lewy Body Parkinson's Disease; Paralysis Agitans; Parkinson's Disease, Idiopathic; Parkinson's Disease, Lewy Body; Primary Parkinsonism
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Radiation: Far Infrared Radiation (5μm to 20μm wavelength)
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Radiation: Far Infrared Radiation (5μm to 20μm wavelength). Far Infrared radiation for 30 to 40 minutes per treatment session.
  Other Names: Far Infrared Radiation

SUMMARY:
Parkinson's disease (PD) is a degenerative disorder of the central nervous system that often impairs the sufferer's motor skills and speech. This study will investigate the use of far infrared radiation to manage, control and treat PD.

DETAILED DESCRIPTION:
Parkinson's disease belongs to a group of conditions called movement disorders. It is characterized by muscle rigidity, tremor, a slowing of physical movement and, in extreme cases, a loss of physical movement. The primary symptoms are the results of decreased stimulation of the motor cortex by the basal ganglia, normally caused by the insufficient formation and action of dopamine, which is produced in the dopaminergic neurons of the brain. PD is both chronic and progressive.

Observations from our research studies indicate that, far infrared rays provide energy to the body, improve the autonomic functions of the nervous system, restore the functions of the endocrine system, strengthen the immune system, improve blood circulation and increase the level of oxygen in the cells and promote the regeneration of muscle cells, nerves and brain cells.

It is hereby postulated that irradiation using far infrared, with wavelength between 5 to 20 microns, of the central nervous system, the endocrine system and the whole body could prevent, control, manage or possibly lead to complete rehabilitation of people who have PD.

ELIGIBILITY:
Inclusion Criteria:

* People with Parkinson's Disease

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Cure for PD | 2 years

SECONDARY OUTCOMES:
Rehabilitation of PD Patients | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada